CLINICAL TRIAL: NCT02045251
Title: AN OPEN-LABEL TRIAL OF REDUCED- DOSE PYLERA (BISMUTH, METRONIDAZOLE, TETRACYCLINE), AMOXICILLIN, AND ESOMEPRAZOLE IN THE TREATMENT OF HELICOBACTER PYLORI INFECTION
Brief Title: An Open-Label Trial Of Reduced- Dose Pylera, Amoxicillin, and Esomeprazole in the Treatment Of Helicobacter Pylori Infection
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unavailability of clarithromycin 250 mg in the market
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM.AS1.33
Record Dates: First submitted 2013-07-18; First posted 2014-01-24 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2013-03

CONDITIONS: Treatment of H. Pylori Infection
Keywords: Helicobacter pylori; H. pylori; Pylera

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional Arm (Experimental): This arm will have 100 patients receiving the proposed Pylera based regimen for 10 days.
  Interventions: Drug: Pylera based reduced regimen

INTERVENTIONS:
Drug: Pylera based reduced regimen — Patients with H. pylori infection will be treated with a 10 day course of reduced Pylera based regimen.

SUMMARY:
Over the years, it has become clear that the first-line triple therapy is losing efficacy worldwide. A capsule containing 3 agents (Pylera®) containing 125mg metronidazole, 140mg bismuth subcitrate potassium, and 125mg tetracycline was made available.

The efficacy of the Pylera capsule was studied in a randomized control trial, in which a quadruple Pylera therapy (Pylera capsule and a PPI) was evaluated against the standard triple regimen. In the study, 3 three-in-one capsules were taken four times daily (after meals and at bedtime).

Given the above, we aim at assessing the effectiveness of fewer pills per day of the Pylera capsule (3 Pylera capsules supplemented with the addition of amoxicillin and esomeprazole twice daily; sum of 10 pills/day for 10 days) in the eradication of H. pylori.

DETAILED DESCRIPTION:
ABSTRACT

Infection with H. pylori has been linked with chronic active gastritis, peptic ulcer disease, adenocarcinoma and Non-Hodgkin's lymphoma of the stomach. Eradication of this organism has been recommended for patients with peptic ulcer disease, low-grade gastric mucosa-associated lymphoid tissue lymphoma, atrophic gastritis, unexplained iron deficiency anemia, chronic idiopathic thrombocytopenic purpura, as well as first-degree relatives of gastric cancer patients. Guidelines still recommend using triple therapy regimen of PPI, clarithromycin and amoxicillin/metronidazole twice daily for 7 to 14 days. Over the years, it has become clear that the first-line triple therapy is losing efficacy worldwide with per protocol (PP) and intent-to-treat (ITT) eradication rates of less than 80%. In light of the low eradication rates of this regimen, quadruple regimens (bismuth and non bismuth based) or alternative fluoroquinolones-based regimens evolved in an attempt to increase the eradication of H. pylori. Most of the new quadruple regimens are clarithromycin-based. Quadruple therapies improved eradication rates to 85-90% but the increasing resistance of H. pylori to clarithromycin rendered the above-mentioned regimens suboptimal. Many attempts to increase the number of antibiotics in treatment regimens were faced with intolerability by patients of the large number of pills and increasing side effects (metallic taste, nausea, etc.). Considering the above, a capsule containing 3 agents (Pylera®) containing 125mg metronidazole, 140mg bismuth subcitrate potassium, and 125mg tetracycline was made available. The importance of such capsule lies in the 3 in 1 packaging and in the avoidance of clarithromycin use and hence the low risk of resistance. The efficacy of the Pylera capsule was studied in a randomized control trial, in which a quadruple Pylera therapy (Pylera capsule and a PPI) was evaluated against the standard triple regimen. In the study, 3 three-in-one capsules were taken four times daily (after meals and at bedtime). An omeprazole capsule was taken with the three single three-in-one capsules after morning and evening meals. Quadruple therapy (Pylera-based) provided superior eradication rates when compared to the standard triple therapy (as high as 80% eradication rate versus 55% on ITT) with similar safety and tolerability [1]. In the aforementioned study, patients on quadruple therapy were taking the sum of 14 pills per day. This big number of pills per day is too high and may threaten compliance and adherence in real life situations outside of controlled clinical trials. This is evidenced by the difference in the PP and ITT eradication rates (93% and 80% respectively) that can be attributed to the load of pill load.

The sensitivity of H. pylori to tetracycline and amoxicillin is very high and resistance is approximately zero [2]. Our local data in Lebanon show essentially no resistance to tetracycline or amoxicillin and a modest rate of metronidazole resistance, similar to Western countries (Fig 1). The use of these antibiotics to treat H. pylori infection is promising. In addition, we have recently shown in 2 separate randomized controlled trials that the reduced or half-dose of antibiotics (including 500 mg bid of amoxicillin and 250 mg bid of metronidazole) can achieve the same eradication of H. pylori at reduced cost and reduced side effects.

Fig 1. In vitro Susceptibility of H. Pylori in Lebanon. Sharara AI, et al. Int J Antimicrob Agents 2000; 19:155-8.

Our studies have shown a declining rate of H. pylori eradication with conventional triple therapy over time (Fig2).

Fig 2. 10-day Legacy Triple Therapy in Lebanon. Soweid A, et al. ACG 2005 [abstract]; Mansour N, et al, Sharara AI. Eur J Gastroenterol Hepatol 2011

Given the above, we aim at assessing the effectiveness of fewer pills per day of the Pylera capsule (3 Pylera capsules supplemented with the addition of amoxicillin and esomeprazole twice daily; sum of 10 pills/day for 10 days) in the eradication of H. pylori. The total dose of drugs is shown in Figure 3.

One hundred patients from the outpatient department and the endoscopy unit at AUBMC will be enrolled in this open-label single arm trial. Patients with positive CLO tests or urea breath tests, or histological documentation of H. pylori infection, will be enrolled in the study. The patients will be followed up by phone calls on day 10 for side effects and for pill count. Patients will be assessed for the presence of these side effects at the end of the treatment (Day 10). A urea breath test will be done for all patients after ≥ 4 weeks of therapy completion and a minimum of 2 weeks of PPI therapy to evaluate eradication rates

Eradication rate will be assessed periodically (every 10 patients) to confirm efficacy with stop points as follows:

Patients 1-10: <60% eradication Patients 1-20: <65% eradication Patients 1-30: <70% eradication Patients 1-40: <75%eradication Patients 1-50: <80% eradication

Fig 3. Doses of drugs of the proposed Pylera regimen compared to the previously studied full-dose and half-dose quadruple (non-bismuth based) regimens.

Study Description:

A- Objective:

The objective of this study is to evaluate the efficacy of the 4 tablets (2 capsules containing metronidazole, bismuth, and tetracycline) plus amoxicillin and esomeprazole) given twice a day for 10 days in the eradication of H. pylori. The primary end point is H. pylori eradication rate on ITT and PP analysis. Secondary endpoints include: (1) tolerability, (2) adverse events of the drug regimen, (3) and cost.

B- Patient population:

One hundred patients from the outpatient department and the endoscopy unit at AUBMC will be enrolled in this open-label trial.

* Inclusion criteria Patients with either positive CLO tests, urea breath tests, or histopathologic documention of H. pylori infection, and agreeing to the study by signing the informed consent.
* Exclusion criteria

  * Age under 18 or older than 80 years
  * Allergies to any of the drugs used
  * Recent antibiotic therapy (within 2 weeks of enrollement)
  * Severe ulcers or bleeding
  * Gastric perforation or obstruction
  * Previous gastrectomy
  * Gastric cancer
  * Pregnancy or lactation
  * Prior eradication therapy for H. pylori
  * Severe concomitant disease or condition making the treatment unlikely to be effective i.e. alcoholism, drug addiction, and history of poor compliance.

C- Design and methods:

After documentation of the H. pylori infection, the primary physician will introduce the patient to the research fellow who will give to the patients a clear explanation of the purpose of the study, risks, and benefits. Those who agree to participate and sign the informed consent will be enrolled in our study. All patients will take the treatment for ten days. The patients will be assessed for side effects on days 5 and 10 of the treatment regimen. The eradication rate will be assessed periodically (every 10 patients for the first 50 patients) for efficacy and the study will be stopped if the target rates are not met. The Pylera tablets will be provided free to patients. However, the amoxicillin and esomeprazole are not provided freely.

Patients will be taking:

* 3 Pylera capsules b.i.d (per capsule: 125mg metronidazole, 125mg tetracycline, 140mg bismuth; i.e. 250mg metronidazole, 250 tetracycline, and 280mg bismuth b.i.d)
* Amoxicillin (Amoxil®) 500 g b.i.d.
* PPI (Esomeprazole 20mg b.i.d)

Compliance and potential side effects will be evaluated by phone calls (day 10) during and shortly after the treatment period. After a minimum of 4 weeks of therapy completion, patients will be asked to present for a urea breath test free of charge in order to evaluate the eradication rate of H. pylori. All patients should be off any PPI for at least two weeks before testing.

D- Statistical Interpretation:

Efficacy of eradication of each group will be evaluated directly from the quotient of the patients with negative urea breath test over the total number of patients enrolled in that group. Success of therapy will be evaluated according to intent-to treat and per-protocol analyses.

ELIGIBILITY:
Inclusion Criteria:

Patients with either positive CLO tests, urea breath tests, or histopathologic documention of H. pylori infection, and agreeing to the study by signing the informed consent.

Exclusion Criteria:

* Age under 18 or older than 80 years
* Allergies to any of the drugs used
* Recent antibiotic therapy (within 2 weeks of enrollement)
* Severe ulcers or bleeding
* Gastric perforation or obstruction
* Previous gastrectomy
* Gastric cancer
* Pregnancy or lactation
* Prior eradication therapy for H. pylori
* Severe concomitant disease or condition making the treatment unlikely to be effective i.e. alcoholism, drug addiction, and history of poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | Eradication
  The rate of eradication of H. pylori using the proposed regimen

SECONDARY OUTCOMES:
Side effects of treatment | Day 10 (at the end of treatment)
  Assessment of side effects of the new regimen

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon